CLINICAL TRIAL: NCT01509287
Title: Metabolic Screening in Patients With Donnai-Barrow Syndrome
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Barbara R. Pober, Principal Investigator and Clinical Geneticist, Massachusetts General Hospital
Other Study IDs: 2009p001589
Record Dates: First submitted 2012-01-10; First posted 2012-01-12 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Donnai-Barrow Syndrome
Keywords: Donnai-Barrow Syndrome (DBS); metabolic testing; genes; genetic
MeSH Terms: conditions — Donnai-Barrow syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, saliva, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Donnai-Barrow Syndrome (DBS): Individuals affected with Donnai-Barrow Syndrome (DBS)
- Unaffected: Healthy family members of individuals affected with Donnai-Barrow Syndrome (DBS)

SUMMARY:
This study focuses on the genetics and metabolism of Donnai-Barrow Syndrome (DBS).

DETAILED DESCRIPTION:
The purpose of this study is to better understand the role of certain nutrients and vitamins in promoting the healthy development of individuals with Donnai-Barrow Syndrome. The investigators hope that the information gained by studying the metabolism of children with Donnai-Barrow Syndrome and their family members will lead to significant advances in the treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

All individuals affected with Donnai-Barrow Syndrome

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children/infants affected with Donnai-Barrow Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2010-03; Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
measures of blood sugar, cholesterol, vitamins A and D, and other compounds | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pober, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States